CLINICAL TRIAL: NCT05825625
Title: Neoadjuvant TiRagolumab, Atezolizumab and Chemotherapy - Dissection of IO Efficacy in NSCLC by Longitudinal tracKing: a Non-randomized, Open-label, Single-arm Phase II Study
Brief Title: NeoTRACK - Dissection of IO Efficacy in NSCLC by Longitudinal tracKing
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Thoraxklinik-Heidelberg gGmbH (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoTRACK; IKF-056 (Other: Institut für Klinische Krebsforschung IKF); 2022-501322-38-00 (Other: EU CT Number)
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; NSCLC; neoadjuvant; surgery; perioperative; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Intervention Model Description: single-arm phase II trial combining chemotherapy with tiragolumab and atezolizumab as neoadjuvant and adjuvant treatment for surgical NSCLC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platinum-based chemotherapy in combination with atezolizumab and tiragolumab (Experimental): Patients will receive 2 cycles of SOC platinum-based chemotherapy as per investigator's choice in combination with atezolizumab and tiragolumab administrated by IV infusion.
  Curative intended surgery will follow after last dose of neoadjuvant treatment. After surgery, patients will receive adjuvant treatment including 2 cycles of platinum-based chemotherapy and atezolizumab plus tiragolumab for up to 1 year. Patients who achieved pCR will receive only atezolizumab plus tiragolumab for up to one year as maintenance therapy.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1,200 mg by IV infusion Q3W.
  Other Names: Tecentriq
Drug: Tiragolumab — Tiragolumab by IV infusion Q3W.
  Other Names: no other name available

SUMMARY:
Prospective, non-randomized, open-label, single-arm phase II trial to investigate the feasibility and efficacy of combining chemotherapy with tiragolumab and atezolizumab as neoadjuvant and adjuvant treatment for surgical NSCLC patients.

DETAILED DESCRIPTION:
The present study is a prospective, investigator-initiated, single-arm, open-label phase II trial. Patients with non-small cell lung cancer of clinical stage II, IIIA and IIIB (T3N2 only) will receive 2 cycles platinum-based standard of care chemotherapy in combination with anti-TIGIT antibody tiragolumab and the anti-PD-L1 antibody atezolizumab followed by curative intent surgery. After surgery, patients not achieving pCR will receive additional 2 cycles chemotherapy in combination with tiragolumab and atezolizumab, followed by tiragolumab/atezolizumab only for up to one year (max 16 cycles) or until intolerable toxicity, disease progression or patients' request, whatever occurs first. Patients with pCR will receive the IO-IO antibodies only (without additional chemotherapy). The objective of this study is to investigate the feasibility, efficacy and safety of combining chemotherapy with tiragolumab and atezolizumab as neoadjuvant and adjuvant treatment for surgical NSCLC patients. Efficacy outcomes will be correlated to the accompanying in-depth translational analyses, which aim to understand the role of the tumor microenvironment in response to IO-IO therapies and to identify biomarkers that may be associated with response and resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Patient* 18 years or older at time of signing informed consent form
3. Histologically confirmed NSCLC of squamous or non-squamous histology
4. Resectable clinical stage II, IIIA and IIIB (T3N2 only) NSCLC (according to UICC 8)
5. Adequate disease staging by PET and/or CT as per SOC (performed ≤ 42 days prior initiation of the study treatment)
6. At least 1 measurable lesion according to RECIST v1.1
7. ECOG performance status ≤ 1
8. Adequate lung and cardiac function for curative intend lung resection (R0) according to German S3 guideline
9. Eligibility to receive a platinum-based neoadjuvant chemotherapy
10. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
11. The patient is willing and able to provide liquid and tissue samples for the accompanying translation project.
12. Adequate bone marrow and renal function including the following:

    * Hemoglobin ≥ 9.0 g/dL
    * Absolute neutrophil count ≥ 1.0 x 109/L
    * Platelets ≥ 75 x 109/L
    * Calculated creatinine clearance ≥ 30 mL/min as determined by the Cockcroft-Gault equation
13. Adequate hepatic function (with stenting for any obstruction, if required) including the following:

    * Serum bilirubin ≤ 3 x institutional upper limit of normal (ULN)
    * AST (SGOT) / ALT (SGPT) and alkaline phosphatase ≤ 2.5x ULN
14. Female patients who are considered as women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
15. Female patients who are considered as WOCBP must use any contraceptive method with a failure rate of less than 1% per year during the treatment as well as up to 5 months after the last dose of IMP. Male patients who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during the treatment as well as at least 5 months after the last dose of IMP. Female patients who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile, see section 5.1.5) as well as azoospermic male patients do not require contraception.

Exclusion Criteria:

1. Treatment in any other clinical trial with an investigational product within 30 days before screening
2. Clinical stage I, IIIB (T4N2), IIIC, nodal NSCLC stage cN3 and stage IV NSCLC
3. Positive testing of activating (TKI-responsive) EGFR-mutation, ROS1-mutation or known ALK fusion oncogene
4. Expected pneumonectomy at baseline to achieve curative intend resection
5. Any concurrent chemotherapy, investigational product (IMP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (e.g. hormone replacement therapy) is acceptable.
6. Malignancies other than NSCLC within 3 years prior to study inclusion with the exception of malignancies with a negligible risk of metastases or death (5-year OS > 90%) like localized prostate cancer, ductal carcinoma in situ, adequately treated carcinoma in situ of the cervix, Stage I uterine cancer, in-situ bladder cancer treated by BCG-Instillation, or non-melanoma skin carcinoma
7. History of allogeneic tissue / solid organ transplant or allogeneic stem cell transplantation
8. History of active primary immunodeficiency.
9. Clinical diagnosis of active tuberculosis.
10. Positive testing for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus (HCV) RNA indicating acute or chronic infection. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
11. Positive testing for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
12. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 5 months after the last dose of atezolizumab/tiragolumab.
13. Active or prior documented autoimmune or inflammatory disorders (including but not limited to diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis, or Wegener's syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto's disease) stable on hormone replacement
    * Patients with controlled Type I diabetes mellitus on an insulin regimen
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
14. Active, uncontrolled inflammatory bowel disease [e.g. ulcerative colitis or Crohn's disease]. Patients in stable remission for more than 1 year may be included.
15. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, interstitial lung disease, gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of atezolizumab/tiragolumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
17. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
18. History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia, drug-induced pneumonitis, or evidence of active pneumonitis on screening chest Computed Tomography (CT) scan.
19. Prior treatment with CD137 agonist or immune checkpoint blockade therapies, such as anti-TIGIT, anti-PD-1 and anti-PD-L1 therapeutic antibody
20. Live vaccine within 30 days prior to first dose of trial treatment
21. Known allergy or hypersensitivity to any component of the chemotherapy regimen or to the IMP or any constituents of the products
22. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
23. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.
24. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
MPR rate after curative intent surgery | 12 weeks
  number of patients with ≤ 10% of residual viable tumor in lung and lymph nodes as evaluated by pathology review, divided by the number of all patients with posttreatment tumor tissue available

SECONDARY OUTCOMES:
Pathological complete response (pCR) | 12 weeks
  Pathological complete response (pCR) is defined as the absence of any viable tumor cells in the entire surgical specimen (resected main lung tumor and resected lymph node tissue).
Radiological response by RECIST v1.1 criteria | 12 weeks
  The radiological response will be assessed according to RECIST v1.1
Event-free survival (EFS) | 78 months
  Event-free survival (EFS) is defined as the time from first dose of the study drug to any of the following events, whichever occurs first: disease progression that precludes surgery, as assessed by the investigator according to RECIST v1.1; local or distant disease recurrence (including occurrence of new primary NSCLC); or death from any cause
Overall survival (OS) | 78 months
  Overall survival is defined as time from treatment initiation (administration of first neoadjuvant cycle) to the date of death from any cause. A subject who has not died at the end of the trial will be censored at last known date alive.
Rate of adverse events and serious adverse events rate | 78 months
  Safety assessments will include physical examinations including performance status (ECOG), clinical laboratory profile and adverse events.
  All observed toxicities and side effects will be graded according to NCI CTCAE v5.0 for all patients and their relationship to the study treatment will be assessed and summarized. The rate of adverse events and serious adverse events rate as well as the frequency of abnormal laboratory parameters will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Florian Eichhorn, Dr., Principal Investigator — Thoraxklinik Heidelberg gGmbH - Universitätsklinikum Heidelberg
Locations (2):
- Germany (2):
  - Universitätsklinikum Essen (AöR)-Westdeutsches Tumorzentrum Essen, Essen
  - Thoraxklinik Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Roesch RM, Schnorbach J, Klotz LV, Griffo R, Thomas M, Stenzinger A, Christopoulos P, Allgaeuer M, Schneider M, Schuler M, Wiesweg M, Schramm A, Bolukbas S, Doerr F, Hegedus B, Cvetkovic J, Kirchner M, Eichhorn ME, Winter H, Bozorgmehr F, Eichhorn F. NeoTRACK trial: Neoadjuvant TiRagolumab, Atezolizumab and Chemotherapy - dissection of IO- efficacy in NSCLC by longitudinal tracKing - protocol of a non-randomised, open-label, single-arm, phase II study. BMJ Open. 2025 Mar 27;15(3):e096617. doi: 10.1136/bmjopen-2024-096617. PMID 40147985